CLINICAL TRIAL: NCT07190534
Title: The Effectiveness of Hydroxychloroquine Versus Methotrexate in the Treatment of Frontal Fibrosing Alopecia in Routine Clinical Care: a Patient Preference Trial
Brief Title: The Effectiveness of Hydroxychloroquine Versus Methotrexate in the Treatment of Frontal Fibrosing Alopecia in Routine Clinical Care: a Patient Preference Trial (FFA Trial)
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Rick Waalboer-Spuij, MD, PhD, Principal Investigator, Erasmus Medical Center
Other Study IDs: 14475
Record Dates: First submitted 2025-09-12; First posted 2025-09-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Frontal Fibrosing Alopecia; Cicatricial Alopecia
Keywords: Frontal fibrosing alopecia; FFA; Cicatricial alopecia; Scarring alopecia; Hair disease; hydroxychloroquine; methotrexate
MeSH Terms: conditions — Alopecia; Hair Diseases | interventions — Hydroxychloroquine; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hydroxychloroquine group: Intervention: hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine (HCQ)
- Methotrexate group: Intervention: methotrexate
  Interventions: Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — 400 mg orally once daily
  Other Names: Plaquenil
  Groups: Hydroxychloroquine group
Drug: Methotrexate (MTX) — 15 mg weekly, orally or subcutaneously (+ concomitant medication: Folic acid 10 mg once weekly, taken 24 hours after MTX)
  Other Names: MTX
  Groups: Methotrexate group

SUMMARY:
Frontal fibrosing alopecia (FFA) is a type of scarring hair loss that mostly affects women and causes permanent hair loss. Two medicines, hydroxychloroquine (HCQ) and methotrexate (MTX), are often used to treat FFA, but it is not yet clear which treatment works better. This study aims to compare the effects of HCQ and MTX in everyday clinical care.

Adults with FFA who choose to start either HCQ or MTX and will be followed for up to 48 weeks.

The main goal is to see how well each medicine helps reduce disease activity, measured by a tool called the Frontal Fibrosing Alopecia Severity Score (FFASS) after 6 months. At each clinic visit, participants will also complete short questionnaires about symptoms, quality of life, and general well-being.

By collecting this information, the study hopes to provide better evidence about how well HCQ and MTX work for FFA, which may help guide future treatment recommendations.

DETAILED DESCRIPTION:
Frontal fibrosing alopecia (FFA) is a form of primary cicatricial alopecia characterized by progressive, irreversible hair loss. It typically affects postmenopausal women. The disease presents with frontotemporal hairline recession, eyebrow loss, and perifollicular inflammation. Although the exact cause remains unclear, an autoimmune-mediated destruction of follicular stem cells is suspected.

Treatment options are limited and largely empirical. Among systemic therapies, hydroxychloroquine (HCQ) and methotrexate (MTX) are the most commonly prescribed in clinical practice. Both drugs are used off-label, and there is no consensus on their effectiveness. Existing studies are mostly retrospective or small-scale. As a result, clinical decision-making is highly variable and evidence-based guidelines are lacking.

This multicenter, prospective patient preference trial has been designed to evaluate the effectiveness of HCQ compared with MTX in adults with FFA under routine clinical care conditions.

Study procedures:

Eligible patients (≥18 years) with a confirmed diagnosis of FFA will be recruited at dermatology outpatient clinics.

Patients will select either HCQ (400 mg daily) or MTX (15 mg weekly, with folate supplementation), according to shared decision-making and standard prescribing protocols.

Follow-up will occur at regular intervals consistent with standard care: baseline, 12, 24, 36, and 48 weeks.

The primary outcome is the change in Frontal Fibrosing Alopecia Severity Score (FFASS) between baseline and 24 weeks. FFASS is a validated composite tool incorporating clinical signs, hairline recession, and patient symptoms.

Secondary outcomes include disease severity across all time points, patient-reported health-related quality of life (Skindex-29, CASIS), adverse events, discontinuation rates, and cost-effectiveness based on health economics instruments (EQ-5D-5L with bolt-ons, ICECAP-A, iMCQ, iPCQ). All FFASS assessments will be performed by two raters using standardized clinical photography and trichoscopy.

Sample size and feasibility:

As FFA is a rare disease, no formal power calculation was performed. Recruitment will continue for 12 months, aiming for a minimum of 25 patients per treatment arm (50 total). This sample size is consistent with exploratory studies in rare conditions and is expected to generate meaningful preliminary evidence.

Statistical analysis:

Analyses will follow the intention-to-treat principle. Primary endpoint comparisons (change in FFASS from baseline to week 24) will be performed using independent-samples tests or non-parametric equivalents, as appropriate. Longitudinal changes will be analyzed with linear mixed-effects models to account for repeated measures and potential confounding factors (e.g., age, sex, disease duration, baseline severity). Because treatment allocation is preference-based rather than randomized, baseline characteristics will be carefully compared and adjusted for in multivariate analyses. Propensity score methods may be applied to further control for allocation bias. Secondary outcomes will be analyzed with similar mixed models or descriptive statistics, depending on variable type.

Data management and quality assurance:

Data will be collected and stored in the validated Castor EDC platform, with patient information pseudonymized. Photos and clinical data will be retained securely for a minimum of 10 years, in line with Erasmus MC guidelines and FAIR data principles (Findable, Accessible, Interoperable, Reusable). Privacy and confidentiality will be strictly maintained, and access will be restricted to authorized research team members.

Risks and burden:

Both HCQ and MTX are well-established systemic treatments in dermatology, prescribed within their standard safety monitoring frameworks. The study does not require additional clinic visits beyond routine care. The only extra element is the completion of short questionnaires, taking approximately 5-15 minutes at specified visits. Risks are therefore considered negligible.

This study addresses an urgent knowledge gap in FFA by providing prospective, systematically collected real-world data on the effectiveness and tolerability of HCQ and MTX. The results are expected to inform future treatment guidelines and improve evidence-based care for this rare and burdensome condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of frontal fibrosing alopecia (FFA)
* Willing and able to provide written informed consent
* Adequate understanding of the Dutch language
* No known contraindications or allergies to hydroxychloroquine (HCQ) or methotrexate (MTX)

Exclusion Criteria:

* Histopathological different diagnosis than FFA.
* Inability to adhere to the study protocol, including medication intake, clinic visits, and questionnaire completion.
* Patients who are ineligible for the HCQ arm (due to contraindications), are automatically included in the MTX arm.

Contraindications HCQ: retinopathy and/or maculopathy/myasthenia gravis/body weight less than 35 kg

- Patients who are ineligible for the MTX arm (due to contraindications), are automatically included in the HCQ arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from dermatology outpatient clinics at Erasmus MC University Medical Center Rotterdam. The study population consists of adults who have been diagnosed with frontal fibrosing alopecia (FFA) during routine clinical care and are considering systemic treatment with hydroxychloroquine or methotrexate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Frontal Fibrosing Alopecia Severity Score (FFASS) change | Baseline to 24 weeks
  The FFASS is a validated scoring system (range 0-25) that captures extent of hairline recession, eyebrow loss, clinical signs of inflammation, and patient symptoms. The primary endpoint is the mean change in FFASS from baseline to 24 weeks, comparing the hydroxychloroquine and methotrexate cohorts.

SECONDARY OUTCOMES:
FFASS change over time | Baseline, Weeks 12, 24, 36, and 48
  Longitudinal change in disease severity as measured by FFASS across all follow-up visits.
Health-Related Quality of Life (HRQoL) | Baseline, Weeks 12, 24, 36, and 48
  Change in patient-reported HRQoL measured by Skindex-29 (dermatology-specific).
Health-Related Quality of Life (HRQoL) | Baseline, Weeks 12, 24, 36, and 48
  Change in patient-reported HRQoL measured by CASIS (hair disease-specific) questionnaire
Adverse Events and Safety | Baseline through Week 48
  Number, type, and severity of adverse events associated with hydroxychloroquine or methotrexate, as reported during routine care monitoring.
Cost-Effectiveness and Health Economic Outcomes | Baseline and Week 24
  Assessment of productivity losses, health care utilization, and broader well-being using EQ-5D-5L
Cost-Effectiveness and Health Economic Outcomes | Baseline and Week 24
  Assessment of productivity losses, health care utilization, and broader well-being using iMCQ/iPCQ
Cost-Effectiveness and Health Economic Outcomes | Baseline and Week 24
  Assessment of productivity losses, health care utilization, and broader well-being using ICECAP-A

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC University Medical Center, Rotterdam, South Holland, Netherlands